CLINICAL TRIAL: NCT01895270
Title: Improving Buprenorphine Detoxification Outcomes With Isradipine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R21DA035325 (NIH); R21DA035325 (NIH)
Record Dates: First submitted 2013-06-25; First posted 2013-07-10 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Opioid Dependence
Keywords: opioid dependence; buprenorphine; isradipine; opioid withdrawal; opioid detoxification
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Isradipine; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isradipine (Experimental): Isradipine controlled-release formulation, 10 mg/day maintenance dose, will be administered according to the following dose procedures: Isradipine ingestion will occur under supervision 6 days per week, and a take-home dose will be given on Saturday for participants to take on Sunday. The initial dose of isradipine or placebo will be given on Day 3 of Week 1. The initial dose of isradipine will be 5 mg/day; the dose will increase to 10 mg/day on Day 3 of Week 3 and will continue through Day 2 of Week 7. On Day 3 of Week 7, isradipine will be decreased to 5 mg/day for 7 days. On Days 3-5 of Week 8, all participants will receive placebo. If ISR side effects are too severe at the 10-mg dose, isradipine will be decreased to 5 mg/day. If ISR side effects are too severe at 5 mg/day, isradipine will be discontinued and the participant will be discharged from the study and referred to local treatment agencies.
  Interventions: Drug: Isradipine
- Placebo (Placebo Comparator): Placebo will consist of microcrystalline cellulose. Two placebo capsules will be administered per day starting week 1 day 3 through the end of the isradipine taper.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Isradipine — Isradipine extended release formulation
  Arms: Isradipine
Drug: Placebo — Placebo will consist of microcrystalline cellulose.
  Other Names: microcrystalline cellulose
  Arms: Placebo

SUMMARY:
This application seeks to address the problem of opioid withdrawal by examining the utility of the L-type calcium channel blocker (CCB) isradipine as an adjunct to BUP detoxification. This project will address the need for improved detoxification strategies by assessing the tolerability and preliminary efficacy of adjunct isradipine during a BUP detoxification in opioid-dependent participants. This pilot clinical trial will determine the potential utility of the L-type CCB isradipine to improve treatment outcomes in up to 60 opioid-dependent individuals undergoing a BUP detoxification procedure. Specifically, this study will determine the efficacy of isradipine to reduce withdrawal symptoms, craving, and illicit use of opioids in opioid-dependent individuals undergoing BUP detoxification and determine the tolerability and safety of controlled-release isradipine (10 mg/day) in opioid-dependent individuals undergoing BUP detoxification. Currently, the only FDA-approved medications for opioid withdrawal are the opioid agonists methadone and BUP, both of which have abuse liability. Our findings, if positive, will support a larger phase II clinical trial.

DETAILED DESCRIPTION:
Opioid dependence continues to be a serious public health problem, particularly with the dramatic rise in prescription opioid abuse. Traditional methods of detoxification from opioids, including tapering off the opioid agonist methadone or buprenorphine (BUP) and supportive treatment of symptomatology with the alpha2-adrenergic receptor agonists, are limited by the high relapse rate and/or lack of efficacy in relieving subjective symptoms. In addition, transitioning individuals from methadone to BUP maintenance has been limited by the need to drastically taper the methadone maintenance dose of methadone-maintained individuals prior to switching to BUP maintenance, which can precipitate opiate withdrawal and relapse. This application takes a novel approach to address the problem of opioid withdrawal by examining the utility of the L-type calcium channel blocker (CCB) isradipine as an adjunct to BUP detoxification. L-type CCBs have been shown to alleviate opioid withdrawal in opioid-treated nonhumans, to be safe and effective in alleviating withdrawal symptoms in human detoxification trials, and to have low abuse potential. Moreover, isradipine was the most effective of several CCBs tested and was more effective than the alpha2-adrenergic agonist clonidine in blocking naloxone-induced behavioral effects without producing self-reported effects associated with high potential for abuse. Thus, this project will address the need for improved detoxification strategies by assessing the tolerability and preliminary efficacy of adjunct isradipine during a BUP detoxification in opioid-dependent participants. The aim of this 8-week randomized, placebo-controlled pilot clinical trial is to determine the potential utility of the L-type CCB isradipine to improve treatment outcomes in up to 60 opioid-dependent individuals undergoing a BUP detoxification procedure. The specific aims are to (Aim 1) determine the efficacy of isradipine to reduce withdrawal symptoms, craving, and illicit use of opioids in opioid-dependent individuals undergoing BUP detoxification and (Aim 2) determine the tolerability and safety of controlled-release isradipine (10 mg/day) in opioid-dependent individuals undergoing BUP detoxification. Currently, the only FDA-approved medications for opioid withdrawal are the opioid agonists methadone and BUP, both of which have abuse liability. Our findings, if positive, will support a larger phase II clinical trial. Ultimately, this work could impact the addiction field by providing another pharmacological tool that is efficacious for treating opioid withdrawal while having minimal abuse liability. This would shift clinical practice, establishing an effective adjunct regimen for BUP detoxification as well as having the potential to enhance transition to naltrexone therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Availability to attend clinic 6 days a week for approximately 30-60 minutes per day.
2. Participants must fulfill DSM-IV criteria for opioid dependence. These criteria will be ascertained in the following manner: the physician will determine whether the individual is appropriate based on several clinical assessments that are routinely employed by methadone program physicians, including history and severity of opioid use, presence of track marks, prior treatment history, self-reported and/or observed signs and symptoms of opioid withdrawal. If any individual's degree of opioid dependence is questionable, that person will be excluded from further consideration as a participant.
3. Participants must submit a urine sample negative for drugs of abuse other than opioids or marijuana prior to starting the study.

Exclusion Criteria:

1. Unstable medical condition or stable medical condition that would interact with study medications or participation.
2. History of major psychiatric disorder (psychosis, schizophrenia, bipolar)
3. Pregnancy or plans to become pregnant or inadequate birth control (adequate birth control includes abstinence, condoms, birth control pills, etc).
4. Present or recent use of over-the-counter psychoactive drug, prescription psychoactive drug or any drug that would have major interaction with drugs to be tested.
5. Liver function tests greater than 3 times normal; BUN and Creatinine outside normal range.
6. EKG abnormalities including but not limited to: bradycardia (<60 bpm); prolonged QTc interval (>450 msec); Wolff-Parkinson White syndrome; wide complex tachycardia; 2nd degree, Mobitz type II heart block; 3rd degree heart block; left or right bundle branch block.
7. Physical dependence on alcohol or drugs other than opioids, marijuana or tobacco (as determined by physician assessment).
8. Pre-existing severe gastrointestinal narrowing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Oliveto, PhD, Principal Investigator — University of Arkansas
Locations (1):
- UAMS Psychiatric Research Institute, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Kumar N, Mancino MJ, Thostenson JD, McGaugh J, Oliveto AH. Feasibility and Preliminary Efficacy of Isradipine During Outpatient Buprenorphine Stabilization and Detoxification: A Pilot Randomized, Placebo-Controlled Trial. Subst Abuse. 2020 Nov 23;14:1178221820970926. doi: 10.1177/1178221820970926. eCollection 2020. PMID 33281447

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 96 consented to screen under a separate screening protocol. Of these, 28 signed consent for this clinical trial. Of 28 signing informed consent, 3 signed informed consent but did not start the trial: one was assigned to ISR and one to PLA. One was lost to follow up before they could be cleared for study entry
Period: Study Medications Induction (W1-4)
Arm/Group | Isradipine | Placebo
Started | 11 | 14
Completed | 5 | 8
Not Completed | 6 | 6
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Vitals outside of ISR dosing parameters | 3 | 2
Not completed — noncompliance- missed medications | 3 | 1
Not completed — Blood pressure issues | 0 | 1
Period: Buprenorphine Taper (W5 to W6D3)
Arm/Group | Isradipine | Placebo
Started | 5 | 7 (1 subject missed meds prior to bup taper so did not start this phase)
Completed | 2 | 2
Not Completed | 3 | 5
Not completed — noncompliance - missed medication | 3 | 5
Period: Isradipine Taper (W7-8)
Arm/Group | Isradipine | Placebo
Started | 2 | 2
Completed | 2 | 0
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: These numbers refer to those that actually started the clinical trial proper.
Groups:
- Total: Total of all reporting groups
Arm/Group | Isradipine | Placebo | Total
Number analyzed (Participants) | 11 | 14 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 14 | 25
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 6 | 10 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 14 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 11 | 13 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 14 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change Over Time in Illicit Opioid Use Via Urine Toxicology Screens During Buprenorphine Taper (Wks 5-6)
Description: Illicit results via urine toxicology screens for heroin and several opioids will be measured thrice weekly during the taper
Time Frame: thrice weekly for approx 2 weeks (taper)
Population: Urine data of subjects that received at least one dose of isradipine and returned for at least one visit in which a urine drug screen was obtained were included in the analysis
Measure: Least Squares Mean (Standard Error); unit: opioid-positive urine
Units Other Than Participants: Urine drug screen results
Arm/Group | Isradipine | Placebo
Number analyzed (Participants) | 5 | 7
Number analyzed (Urine drug screen results) | 7 | 7
opioid-positive urine | -1.25 (0.74) | -0.36 (0.58)
Statistical Analysis 1: Comparison: Isradipine vs Placebo; Test type: Superiority; p = .42, Mixed Models Analysis; Slope = .34, Standard Error of Mean .42

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Participants were queried about their symptoms at every visit and a symptoms form was completed. If the symptom had not been experienced before or was at a greater intensity than experienced previously, then it was considered an adverse event.
Arm/Group | Isradipine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/14
Other Adverse Events (participants affected / at risk) | 10/11 | 8/14
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isradipine (N=11) | Placebo (N=14)
Flushing (Vascular disorders) | 3 (3) | 2 (3)
Headache (Vascular disorders) | 4 (4) | 2 (3)
lethargy, drowsiness, sleepiness, tired (General disorders) | 4 (4) | 4 (5)
vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Tingling, burning in upper extremities (Nervous system disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Itchy bug bite(s) (General disorders) | 2 (2) | 0 (0)
abdominal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
swelling in extremities (Vascular disorders) | 4 (4) | 0 (0)
Change in urine color (Renal and urinary disorders) | 2 (2) | 0 (0)
Increased urination (Renal and urinary disorders) | 2 (2) | 3 (3)
Night sweats/sweating (General disorders) | 0 (0) | 2 (2)
Dizziness, Lightheadedness (Vascular disorders) | 2 (2) | 1 (1)
constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
Results are limited by the high dropout rate. Because opioid dependent individuals tend to have relatively low pressure, the feasibility of using an immediate-formulation of a calcium channel blocker is unclear.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No